CLINICAL TRIAL: NCT06727799
Title: A Non-Treatment Clinical Evaluation of the ELITA Single Piece Patient Interface (PI) for Docking Procedure With the ELITA System
Brief Title: A Non-Treatment Clinical Evaluation of the ELITA Single Piece Patient Interface for Docking Procedure With the ELITA
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CHTA110SDOK
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Diagnostic Test: One eye of each subject will have corneal marks placed and will be docked at the study visit.
  Interventions: Diagnostic Test: Docking Assessment / Observation

INTERVENTIONS:
Diagnostic Test: Docking Assessment / Observation — One eye of each subject will have corneal marks placed and will be docked at the study visit.

SUMMARY:
Open label, prospective, randomized, multicenter, measurement only feasibility study to evaluate the docking procedure using the ELITA Single Piece Patient interface in conjunction with the ELITA system

ELIGIBILITY:
Inclusion Criteria: All criteria apply to both eyes:

* Minimum 22 years of age at the time the informed consent form is signed
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the USA/State
* Ability to understand and respond to a questionnaire in English

Exclusion Criteria: All criteria apply to both eyes:

* History of prior corneal refractive surgery (LASIK, LASEK, RK, PRK, SMILE, etc.), intraocular surgery, cataract extraction or corneal transplant surgery (DSEK, DMEK, DALK, PKP, etc.)

  * History of corneal abnormalities such as stromal, epithelial, or endothelial dystrophies or retinal abnormalities, retinal degeneration or other abnormalities
  * Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
  * History of or active ophthalmic disease or abnormality (including, but not limited to, symptomatic blepharitis, recurrent corneal erosion, clinically significant dry eye syndrome or symptoms, neovascularization > 1 mm from limbus), retinal detachment/repair (including but not limited to any curative or preventative laser treatment of holes, tears, or lattice degeneration), clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm and visible on topography, at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma
  * Ocular hypertension (IOP > 21 mmHg), glaucoma, glaucoma suspect, or subjects taking any medication for these conditions
  * Any abnormality of the optic nerve or vasculature by history or direct evaluation
  * History or current diagnosis of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity, or control, will specifically exclude subjects from eligibility.

Subjects with active ocular infection

* Use of systemic or ocular medications that may affect vision
* Known sensitivity or inappropriate responsiveness to any of the medications used in the study Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.) History or presence of amblyopia
* Concurrent participation or participation in an interventional (i.e., surgical or pharmaceutical interventional) clinical trial within 14 days prior to the 1st study visit.

Subject who is known to be pregnant or breast feeding

• Subjects who belong to vulnerable populations, including but not limited to minors, pregnant individuals, individuals with cognitive impairments, employees of the clinical site or JJV and their immediate family members (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse), individuals unable to provide inform consent, and those who may be subject to coercion or undue influence

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During the evaluation phase, approximately 50 eyes, with a minimum of 20 eyes of East Asian descent (based on demographics) will be enrolled.
  During the confirmation phase, approximately 50 eyes, with a minimum of 20 eyes of East Asian descent (based on demographics) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Successful Docking of Single PI using ELITA | 1 month
  Applanation of the cornea with the Patient interface resulting meniscus formation at PI interface of at least 10 mm in diameter with continuous vacuum suction engaged and no observed eye movement upon successful vacuum engagement that allows centration of a 9 mm flap based on GUI overlay on the centration screen

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford Eye Laser Center, Palo Alto, California
  - Hoopes Vision, Draper, Utah

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu